CLINICAL TRIAL: NCT03872596
Title: A Phase 1, 2-Part, Open-Label, Randomized, Crossover Pilot Trial to Assess the Relative Bioavailability of Quetiapine Versus Seroquel® 300-mg Oral Tablets in Subjects With Schizophrenia or Bipolar Disorder and 25-mg Oral Tablets in Healthy Subjects
Brief Title: Trial to Assess the Bioavailability of Quetiapine Versus Seroquel® in Subjects With Schizophrenia or Bipolar Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 304-201-00001
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-06

CONDITIONS: Bipolar Disorder; Schizophrenia
Keywords: Seroquel; Digital Medicine Quetiapine; Pharmacokinetics; Bioavailability
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Intervention Model Description: This is a two-part, crossover study. In Part A, participants will be randomized into one of three treatment sequences, each receiving Seroquel immediate release (IR) 300mg, Quetiapine Formulation A 300mg and Quetiapine Formulation B 300mg. In Part B, participants will be randomized into one of two treatment sequences, each receiving Seroquel IR 25mg and Quetiapine 25mg, the formulation of which will be established in Part A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part A: Sequence 1 (Experimental): Titration Period:
  All participants will complete the titration period to establish tolerability. Depending on exposure prior to the trial, participants will titrate up to and including a dose of 300mg twice a day (BID) prior to randomization.
  Treatment Period:
  Participants will receive Seroquel IR (tablet, orally, 300mg, BID) on Days 1-5, Quetiapine Formulation A (tablet, orally, 300mg, BID) on Days 6-10 and Quetiapine Formulation B (tablet, orally, 300mg, BID) on Days 11-15.
  Interventions: Drug: Seroquel IR 300mg; Drug: Quetiapine Formulation A 300mg; Drug: Quetiapine Formulation B 300mg
- Part A: Sequence 2 (Experimental): Titration Period:
  All participants will complete the titration period to establish tolerability. Depending on exposure prior to the trial, participants will titrate up to and including a dose of 300mg BID prior to randomization.
  Treatment Period:
  Participants will receive Quetiapine Formulation A (tablet, orally, 300mg, BID) on Days 1-5, Quetiapine Formulation B (tablet, orally, 300mg, BID) on Days 6-10 and Seroquel IR (tablet, orally, 300mg, BID) on Days 11-15.
  Interventions: Drug: Seroquel IR 300mg; Drug: Quetiapine Formulation A 300mg; Drug: Quetiapine Formulation B 300mg
- Part A: Sequence 3 (Experimental): Titration Period:
  All participants will complete the titration period to establish tolerability. Depending on exposure prior to the trial, participants will titrate up to and including a dose of 300mg BID prior to randomization.
  Treatment Period:
  Participants will receive Quetiapine Formulation B (tablet, orally, 300mg, BID) on Days 1-5, Seroquel IR (tablet, orally, 300mg, BID) on Days 6-10 and Quetiapine Formulation A (tablet, orally, 300mg, BID) on Days 11-15.
  Interventions: Drug: Seroquel IR 300mg; Drug: Quetiapine Formulation A 300mg; Drug: Quetiapine Formulation B 300mg
- Part B: Sequence 1 (Experimental): Participants will receive Seroquel IR (tablet, orally, 25mg) on Day 1 and Quetiapine formulation established in Part A (tablet, orally, 25mg) on Day 4.
  Interventions: Drug: Seroquel IR 25mg; Drug: Quetiapine Formulation 25mg
- Part B: Sequence 2 (Experimental): Participants will receive Quetiapine formulation established in Part A (tablet, orally, 25mg) on Day 1 and Seroquel IR (tablet, orally, 25mg) on Day 4.
  Interventions: Drug: Seroquel IR 25mg; Drug: Quetiapine Formulation 25mg

INTERVENTIONS:
Drug: Seroquel IR 300mg — Administered during Part A, administered orally BID with water, over 5 days.
  Arms: Part A: Sequence 1; Part A: Sequence 2; Part A: Sequence 3
Drug: Seroquel IR 25mg — Administered during Part B, as a single, 25mg dose taken with water.
  Arms: Part B: Sequence 1; Part B: Sequence 2
Drug: Quetiapine Formulation A 300mg — Administered during Part A, administered orally BID with water, over 5 days.
  Arms: Part A: Sequence 1; Part A: Sequence 2; Part A: Sequence 3
Drug: Quetiapine Formulation B 300mg — Administered during Part A, administered orally BID with water, over 5 days.
  Arms: Part A: Sequence 1; Part A: Sequence 2; Part A: Sequence 3
Drug: Quetiapine Formulation 25mg — Administered during Part B, as a single, 25mg dose taken with water.
  Arms: Part B: Sequence 1; Part B: Sequence 2

SUMMARY:
This is a two-part trial.

The primary objective of Part A is to estimate the ratio of geometric means of pharmacokinetic (PK) parameters and their within-subject variability for the 300mg quetiapine tablet formulation A and the 300mg quetiapine tablet formulation B compared to 300mg Seroquel.

The primary objective of Part B is to estimate the ratio of geometric means of PK parameters and their within-subject variability for the selected tablet formulation from Part A of 25mg quetiapine compared to 25mg Seroquel.

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Must have a current diagnosis of schizophrenia or bipolar disorder, as determined by the Diagnostic and Statistical Manual of Mental Disorders Version 5 (DSM-5) criteria.
* Must have a Body Mass Index between 18 and 35 kg/m^2.
* Good physical health as determined by no clinically significant deviation from normal, in the opinion of the investigator, in medical history, clinical laboratory determination, ECGs, or physical examinations.
* Participants must be considered stable, per the investigator's judgment, on one of the following atypical oral antipsychotic medications at an adequate dose (eg, low- to mid-range of the recommended dose range for the treatment of schizophrenia or bipolar disorder, according to the manufacturer labeling) and for an adequate duration (30 days) prior to the administration of IMP: aripiprazole, brexpiprazole, risperidone, olanzapine, quetiapine, ziprasidone, paliperidone, cariprazine, lurasidone, and asenapine. Other oral antipsychotic medications may be allowed if approved by the medical monitor and sponsor; however, clozapine will not be allowed. Per the investigator's judgment, they should be comfortable with the participant discontinuing background antipsychotic therapy during the trial period and then restarting the antipsychotic therapy once trial participation has been completed.

Part B:

* Male or female participants between 18 and 45 years of age, inclusive.
* Must have a Body Mass Index between 18 and 32 kg/m^2.
* Good physical health as determined by no clinically significant deviation from normal, in the opinion of the investigator, in medical history, clinical laboratory determination, ECGs, or physical examinations.
* Able to provide informed consent prior to the initiation of any protocol-related procedures.
* Male and female participants who are surgically sterile, female participants who have been postmenopausal for at least 12 consecutive months prior to the screening visit, or male participants/female participants (of childbearing potential) who agree to practice 2 of the approved birth control methods from the screening visit and for at least 30 days after the last dose of IMP for a female participant or 80 days after the last dose of IMP for a male participant.

Exclusion Criteria:

Part A:

* Participants who are unable to stop receiving varenicline beyond the screening visit. If a participant is receiving varenicline at the screening visit, attempts should be made to discontinue the medication, if clinically feasible, to allow potential participants to enter the trial.
* Participants who have a significant risk of committing suicide based on history, routine psychiatric status examination, investigator's judgment, or who have an answer of "yes" on questions 4 or 5 (current or over the last 3 months) on the Baseline/Screening Version of the C-SSRS or participants with any suicidal behavior during the 6 months prior to the screening visit.
* Participants currently in an acute relapse of schizophrenia as assessed by the investigator. Bipolar participants who currently have an unstable mood (manic, mixed, or depressed) as assessed by the investigator.
* Participants with a current DSM-5 diagnosis other than schizophrenia or bipolar disorder, including schizoaffective disorder, major depressive disorder, delirium, dementia, amnestic, or other cognitive disorders. Also, participants with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Use of any moderate-strong CYP3A4 inhibitor or inducer within 14 days or 5 plasma half-lives (whichever is longer) prior to the administration of IMP and for the duration of the trial. Weak CYP3A4 inhibitors, including valproic acid, may be allowed based on the investigator's judgment, provided the participant has been on a stable dose for at least 30 days prior to IMP administration and throughout the duration of the trial.
* Participants with a history of neuroleptic malignant syndrome, seizure disorder, or clinically significant tardive dyskinesia as assessed by the investigator.
* Subjects with a history of any significant drug allergy or known or suspected hypersensitivity to antipsychotics, in particular to quetiapine.
* Participants who are maintained on long-acting insulin.
* Any participant who does not successfully tolerate a quetiapine dose of 300 mg BID during the titration period of this trial.

Part B:

* History of any significant drug allergy to quetiapine, prescription drugs, non-prescription drugs, or food.
* Any history of significant bleeding or hemorrhagic tendencies.
* Exposure to any substances known to stimulate hepatic microsomal enzymes within 30 days prior to screening through the end of the trial (eg, occupational exposure to pesticides, organic solvents, etc).
* Participants who have supine blood pressure after resting for ≥ 5 minutes, higher than 130/80 mmHg or lower than 100/50 mmHg (systolic/diastolic). The sponsor may allow exceptions if they are not deemed clinically significant.
* Participants who have a supine pulse rate, after resting for ≥ 5 minutes, outside the range of 60 to 90 beats per minute. The sponsor may allow exceptions if they are not deemed clinically significant (eg, bradycardia attributable to superior physical fitness).
* History of serious mental disorders that, in the opinion of the investigator, would exclude the participant from participating in this trial.
* Use of any CYP3A4 inhibitors or CYP3A4 inducers within 14 days or 5 plasma half-lives (whichever is longer) prior to the administration of IMP and for the duration of the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) for Quetiapine | Pre-dose on days 4, 9 and 14, 12 hours post morning dose on Days 4, 9 and 14 and pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 3, 4, 6, 8, 10 and 12 hours post morning dose on days 5, 10 and 15
  Pharmacokinetic endpoint analysis will be done separately for formulation A and formulation B.
Part A: Area Under the Concentration-Time Curve Calculated to the Last Observable Concentration at Time t (AUCt) for Quetiapine | Pre-dose on days 4, 9 and 14, 12 hours post morning dose on Days 4, 9 and 14 and pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 3, 4, 6, 8, 10 and 12 hours post morning dose on days 5, 10 and 15
  Pharmacokinetic endpoint analysis will be done separately for formulation A and formulation B.
Part B: Maximum Observed Plasma Concentration (Cmax) for Quetiapine | Predose (within 30 minutes prior to dosing), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12 (Days 1 to 4), 24, 36 (Days 2 and 5), and 48 (Days 3 and 6) hours post dose
Part B: Area Under the Concentration-Time Curve Calculated to the Last Observable Concentration at Time t (AUCt) for Quetiapine | Predose (within 30 minutes prior to dosing), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12 (Days 1 to 4), 24, 36 (Days 2 and 5), and 48 (Days 3 and 6) hours post dose
Part B: Area Under the Concentration-Time Curve from Time Zero to Infinity (AUC∞) for Quetiapine | Predose (within 30 minutes prior to dosing), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12 (Days 1 to 4), 24, 36 (Days 2 and 5), and 48 (Days 3 and 6) hours post dose

SECONDARY OUTCOMES:
Part A: Time to Maximum (Peak) Plasma Concentration (tmax) for Quetiapine | Pre-dose on days 4, 9 and 14, 12 hours post morning dose on Days 4, 9 and 14 and pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 3, 4, 6, 8, 10 and 12 hours post morning dose on days 5, 10 and 15
  Pharmacokinetic endpoint analysis will be done separately for formulation A and formulation B.
Part A: Terminal-Phase Elimination Half-Life (t1/2,z) for Quetiapine | Pre-dose on days 4, 9 and 14, 12 hours post morning dose on Days 4, 9 and 14 and pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 3, 4, 6, 8, 10 and 12 hours post morning dose on days 5, 10 and 15
  Pharmacokinetic endpoint analysis will be done separately for formulation A and formulation B.
Part A: Apparent Clearance of Drug from Plasma After Extravascular Administration (CL/F) for Quetiapine | Pre-dose on days 4, 9 and 14, 12 hours post morning dose on Days 4, 9 and 14 and pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 3, 4, 6, 8, 10 and 12 hours post morning dose on days 5, 10 and 15
  Pharmacokinetic endpoint analysis will be done separately for formulation A and formulation B.
Part A: Percentage of Participants who Experience at Least One Treatment-Emergent Adverse Event | Day 1 to End of Follow-Up (Day 45[+/- 2 days])
  An adverse event is defined as as any untoward medical occurrence in a clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. A Treatment-Emergent Adverse Event (TEAE) is defined as an adverse event that occurs after treatment has begun.
Part A: Percentage of Participants who Experience a Clinically Significant Change from Baseline in Vital Signs | Baseline (Day -1) to Day 11
  Vital signs will include blood pressure, heart rate, temperature, and respiratory rate.
Part A: Percentage of Participants who Experience a Significant Change from Baseline in ECGs | Baseline (Day -1) to Day 11
  Standard 12-lead electrocardiograms will be used.
Part A: Percentage of Participants who Experience a Significant Change from Baseline in Clinical Laboratory Tests | Baseline (Day -1) to Day 15
  Clinical laboratory tests will be conducted at scheduled time points during Part A and Part B, including hematology, urinalysis, serum chemistry, drug screen and additional tests.
Part A: Change from Baseline in Columbia-Suicide Severity Rating Scale Score | Baseline (Day -1) and Day 15
  Suicidality will be monitored throughout the trial using the C-SSRS (Columbia-Suicide Severity Rating Scale). This scale consists of a baseline evaluation that assesses the lifetime experience of the subject with suicide events and suicidal ideation and a post-baseline evaluation that focuses on suicidality since the last assessment.The Baseline/ Screening Version and the Since Last Visit version of the C-SSRS will be completed by trained trial site staff at each visit. A numerical score will correspond to one of ten categories relating to suicidal ideation and suicidal behavior. A higher score indicates a higher risk of suicidal behavior, but an answer of 'yes' to any question indicates some risk.
Part B: Time to Maximum (Peak) Plasma Concentration (tmax) for Quetiapine | Predose (within 30 minutes prior to dosing), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12 (Days 1 to 4), 24, 36 (Days 2 and 5), and 48 (Days 3 and 6) hours post dose
Part B: Terminal-Phase Elimination Half-Life (t1/2,z) for Quetiapine | Predose (within 30 minutes prior to dosing), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12 (Days 1 to 4), 24, 36 (Days 2 and 5), and 48 (Days 3 and 6) hours post dose
Part B: Apparent Clearance of Drug from Plasma After Extravascular Administration (CL/F) for Quetiapine | Predose (within 30 minutes prior to dosing), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12 (Days 1 to 4), 24, 36 (Days 2 and 5), and 48 (Days 3 and 6) hours post dose
Part B: Percentage of Participants who Experience at Least One Treatment-Emergent Adverse Event | Day 1 to End of Follow-Up (Day 34 [+ 2 Days])
  An adverse event is defined as as any untoward medical occurrence in a clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. A Treatment-Emergent Adverse Event (TEAE) is defined as an adverse event that occurs after treatment has begun.
Part B: Percentage of Participants who Experience a Clinically Significant Change from Baseline in Vital Signs | Baseline (Day -1) to Day 6
Part B: Percentage of Participants who Experience a Significant Change from Baseline in ECGs | Baseline (Day -1) to Day 6
  Standard 12-lead electrocardiograms will be used.
Part B: Percentage of Participants who Experience a Significant Change from Baseline in Clinical Laboratory Tests | Baseline (Day -1) to Day 6
  Clinical laboratory tests will be conducted at scheduled time points during Part A and Part B, including hematology, urinalysis, serum chemistry, drug screen and additional tests.
Part B: Change from Baseline in Columbia-Suicide Severity Rating Scale Score | Baseline (Day -1) and Day 6
  Suicidality will be monitored throughout the trial using the C-SSRS (Columbia-Suicide Severity Rating Scale). This scale consists of a baseline evaluation that assesses the lifetime experience of the subject with suicide events and suicidal ideation and a post-baseline evaluation that focuses on suicidality since the last assessment.The Baseline/ Screening Version and the Since Last Visit version of the C-SSRS will be completed by trained trial site staff at each visit. A numerical score will correspond to one of ten categories relating to suicidal ideation and suicidal behavior. A higher score indicates a higher risk of suicidal behavior, but an answer of 'yes' to any question indicates some risk.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Roos, M.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (1):
- Collaborative Neurosciences Network, LLC, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com